CLINICAL TRIAL: NCT03935997
Title: Implementing, Evaluating, and Scaling Up of the Strengthening a Palliative Approach in Long Term Care (SPA-LTC) Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Alberta Health services (Other); Hospice Palliative Care Ontario (Unknown); Canadian Hospice Palliative Care Association (Unknown); Canadian Virtual Hospice (Unknown); Saskatchewan Health Authority - Regina Area (Other); Interlake-Eastern Regional Health Authority (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SPA-LTC408466
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-11

CONDITIONS: Frail Elderly Syndrome
Keywords: Palliative care; End of life care; Long-term care; Nursing home
MeSH Terms: interventions — Long-Term Care

STUDY DESIGN:
Intervention Model Description: Within each of the three provinces, six LTC homes will be randomly selected, and then randomly allocated using a 1:1 ratio, stratified according to province, to either the intervention or control group using a computer-generated list. For each province, three LTC homes will receive the intervention and three will receive usual care. A biostatistician not involved in recruitment will generate group assignments.
Masking Description: There is no need to mask participants, clinicians or research staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Within the intervention arm 9 long-term care homes will receive the SPA-LTC program:3 in Ontario; 3 in Saskatchewan and 3 in Manitoba.
  Interventions: Other: Strengthening a Palliative Approach in Long-Term Care (SPA-LTC) Program
- Control (No Intervention): Within the control arm 9 long-term care homes will receive the standard of care: 3 in Ontario; 3 in Saskatchewan and 3 in Manitoba.

INTERVENTIONS:
Other: Strengthening a Palliative Approach in Long-Term Care (SPA-LTC) Program — Our team will work with long-term care homes in the study to implement the Strengthening a Palliative Approach in Long Term Care (SPA-LTC) which consists of the following core, evidence-informed components:
  Palliative Champion Teams (to provide leadership and support implementation); Palliative Care Education (including illness trajectory pamphlets); Comfort Care Rounds with staff (for capacity building and reflection); Prognostic Tools to trigger end-of-life discussions; Palliative Care Conferences with families and residents; Bereavement Pamphlets; and Post-Bereavement Follow-Up for families, and staff.
  Arms: Intervention

SUMMARY:
This study will evaluate the implementation of the Strengthening a Palliative Approach in Long-Term Care (SPA-LTC) program using a cross-jurisdictional, effectiveness-implementation type II hybrid design (dual testing of clinical and implementation interventions) to assess the implementation (feasibility, fidelity, reach, sustainability) and effectiveness (family satisfaction, staff knowledge and confidence implementing a palliative approach to care, hospital use).

DETAILED DESCRIPTION:
The SPA-LTC program has been developed and refined through prior participatory action based studies.

Evidence-based components of the program include:

Palliative Champion Teams; Palliative Care Education, including illness-trajectory pamphlets for staff and family members; Comfort Care Rounds with staff; Prognostic Tools to trigger end-of-life discussions; Palliative Care Conferences; Bereavement Pamphlets for families; and Post-Bereavement Follow-Up for families, and staff

The goal is to implement and assess this program across three provinces in Canada (Ontario, Saskatchewan, Manitoba). The investigators will use the findings to revise the program and inform the scaling up of the program across diverse settings and provinces.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking LTC residents with a score of 50% or less on the Palliative Performance Scale.

Exclusion Criteria:

* Non-English speaking LTC residents
* residents with a score of more than 50% on the Palliative Performance Scale.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Emergency Department Visits in the Resident's Last Year of Life | All residents in the home who died one year prior to the implementation and one year prior to the date of death for all residents in the home who die during the study intervention period.

SECONDARY OUTCOMES:
Family Perceptions of End of Life Care | Survey completed at enrolment into the study; survey completed 2 months after the Family Care Conference or 1 month after the end of the intervention period if no Family Care Conference occurred.
  Survey
Family Experiences with End of Life Care | Interview completed at enrolment into the study; survey completed 2 months after the Family Care Conference or 1 month after the end of the intervention period if no Family Care Conference occurred.
  Interview
Staff Knowledge about a Palliative Approach to Care | All staff in all participating long-term care homes will complete a staff survey at 2 points in the study: at the beginning and the end of the intervention
  Survey
Number of Hospital Transfers per Resident | Chart audit at start of the trial to capture data on residents who died in the year prior to the trial. Chart audits also during the transition phase prior to Steps 2 and 3; and one month after the intervention period for the trial ends.
  Chart data at each study site will be audited to capture data on the number of hospital transfers in the last year of life for residents who died 1 year before the trial or who die during the trial.
Number of Hospital Deaths during the trial | Chart audit at start of the trial to capture data on residents who died in the year prior to the trial. Chart audits also during the transition phase prior to Steps 2 and 3; and one month after the intervention period for the trial ends.
  Chart data at each study site will be audited to capture data on the number of hospital deaths in the year prior to the trial and during the trial.
  Chart data at each study site will be audited to capture data on the number of hospital transfers in the residents last year of life.
Bereaved Family Satisfaction with End of Life Care | 6 weeks to 2 months after the resident's death
  Qualitative interview with family members whose loved one died during the trial.
Resident Satisfaction with End of Life Care | At the time of enrolment and 2 months after the Family Care Conference or 1 month after the intervention period if no Family Care Conference occurred.
  Qualitative interview with residents who are enrolled in the trial

OTHER OUTCOMES:
Fidelity of the Intervention | Checklist completed weekly during the intervention period for up to 160 weeks.
  Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Kaasalainen, PhD, Principal Investigator — McMaster University, School of Nursing
Locations (4):
- Canada (4):
  - University of Manitoba, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - University of Regina, Regina, Saskatchewan
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Sussman T, Kaasalainen S, Lee E, Akhtar-Danesh N, Strachan PH, Brazil K, Bonifas R, Bourgeois-Guerin V, Durivage P, Papaioannou A, Young L. Condition-Specific Pamphlets to Improve End-of-life Communication in Long-term Care: Staff Perceptions on Usability and Use. J Am Med Dir Assoc. 2019 Mar;20(3):262-267. doi: 10.1016/j.jamda.2018.11.009. Epub 2018 Dec 21. PMID 30583908
- [Background] Thompson G, Shindruk C, Wickson-Griffiths A, Sussman T, Hunter P, McClement S, Chochinov H, McCleary L, Kaasalainen S, Venturato L. "Who would want to die like that?" Perspectives on dying alone in a long-term care setting. Death Stud. 2019;43(8):509-520. doi: 10.1080/07481187.2018.1491484. Epub 2018 Sep 12. PMID 30207512
- [Background] Sussman T, Kaasalainen S, Bui M, Akhtar-Danesh N, Mintzberg S, Strachan P. "Now I Don't Have to Guess": Using Pamphlets to Encourage Residents and Families/Friends to Engage in Advance Care Planning in Long-Term Care. Gerontol Geriatr Med. 2017 Dec 20;3:2333721417747323. doi: 10.1177/2333721417747323. eCollection 2017 Jan-Dec. PMID 29308424
- [Background] Durepos P, Kaasalainen S, Sussman T, Parker D, Brazil K, Mintzberg S, Te A. Family care conferences in long-term care: Exploring content and processes in end-of-life communication. Palliat Support Care. 2018 Oct;16(5):590-601. doi: 10.1017/S1478951517000773. Epub 2017 Dec 29. PMID 29284551
- [Background] Kaasalainen S, Sussman T, Durepos P, McCleary L, Ploeg J, Thompson G; SPA-LTC Team. What Are Staff Perceptions About Their Current Use of Emergency Departments for Long-Term Care Residents at End of Life? Clin Nurs Res. 2019 Jul;28(6):692-707. doi: 10.1177/1054773817749125. Epub 2017 Dec 22. PMID 29271241
- See also: SPA-LTC webpage (housed on the Canadian Hospice Palliative Care Association website) — http://www.chpca.net/projects-and-advocacy/projects/strengthening-a-palliative-approach-in-long-term-care-spa-ltc-project/spa-ltc-model.aspx